CLINICAL TRIAL: NCT04688983
Title: An Open Label, 3-arm, Randomised Phase II Study to Compare the Safety and Efficacy of Ponatinib in Combination With Either Chemotherapy or Blinatumomab With Imatinib Plus Chemotherapy as Front-line Therapy for Patients Aged 55 Years and Over With Philadelphia Chromosome Positive (Ph+ or BCR-ABL+) Acute Lymphoblastic Leukemia (ALL)
Brief Title: Study in Adult Ph-positive ALL
Acronym: EWALL-Ph-03
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cardiff University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SPON-1751-19
Record Dates: First submitted 2020-12-17; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Acute Lymphoblastic Leukemia, Adult
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — ponatinib; blinatumomab; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Active Comparator): Ponatinib plus standard induction and consolidation
  Interventions: Drug: Ponatinib
- Arm 2 (Active Comparator): Imatinib plus standard induction and consolidation (comparator arm)
  Interventions: Drug: Imatinib
- Arm 3 (Experimental): Ponatinib plus Blinatumomab
  Interventions: Drug: Ponatinib; Drug: Blinatumomab

INTERVENTIONS:
Drug: Ponatinib — 30 mg QD starting day 1, given continuously unless interruption required for toxicity
  Arms: Arm 1; Arm 3
Drug: Blinatumomab — A single cycle of blinatumomab treatment is 6 weeks in duration, which includes 4 weeks of blinatumomab CIVI followed by a 2-week treatment-free interval.
  Other Names: Blincyto
  Arms: Arm 3
Drug: Imatinib — starting day 1, given orally at 400mg BID continuously for 8 weeks
  Arms: Arm 2

SUMMARY:
An Open Label, 3-arm, Randomised Phase II Study to Compare the Safety and Efficacy of Ponatinib in Combination With Either Chemotherapy or Blinatumomab With Imatinib Plus Chemotherapy as Front-line Therapy for Patients Aged 55 Years and Over With Philadelphia Chromosome Positive (Ph+ or BCR-ABL+) Acute Lymphoblastic Leukemia (ALL)

DETAILED DESCRIPTION:
Acute lymphoblastic leukemia (ALL) develops when a certain type of immature bone marrow cell called a lymphoblast becomes malignant, resulting in uncontrolled growth and suppression of normal blood cell development. Leukemic blast cells accumulate in the bone marrow and blood and may involve other organs such as the central nervous system (CNS). The most frequent subtype of ALL observed in adults is caused by a genetic aberration called a Philadelphia (Ph) chromosome and is thus referred to as Ph+ ALL. In this type of ALL, a gene called BCR and a gene called ABL are fused by a process known as translocation. This leads to formation of an atypical gene called BCR-ABL and formation of a protein known as the BCR-ABL oncoprotein. This protein, a so-called tyrosine kinase, activates and disrupts many signaling pathways in the cell and is directly responsible for the development of Ph+ ALL, which is one of the most aggressive types of leukaemia.

Treatment options for Ph+ ALL were much improved by a family of drugs called tyrosine kinase inhibitors (TKI), which bind to - and block the activity of - the BCR-ABL kinase. The first of these drugs to be developed is called imatinib (brand name glivec), which has become a standard component of therapy for Ph+ ALL worldwide, usually combined with steroids and/or cytotoxic chemotherapy typically used for ALL. In the vast majority of patients, this treatment is initially able to reduce the burden of the disease to a very low level (complete remission). Unfortunately, the leukemic cells eventually become resistant to imatinib, causing the disease to reappear (relapse). A commonly observed mechanism of resistance to TKI is the development of mutations in the BCR-ABL gene, as a result of which the drug can no longer bind to the kinase, leading to its reactivation. For this reason, stem cell transplantation from a sibling or unrelated donor is considered the most effective treatment to achieve cure.

In the last couple of years, 2nd generation TKI (Dasatinib and Nilotinib) which are more active than imatinib have been tested in clinical trials in patients with Ph+ ALL. Although these newer TKI show activity towards mutated BCR-ABL not inhibited by imatinib, the same basic mechanisms of resistance apply to these drugs, and they have not been shown to result in substantially longer survival than imatinib. In particular, a BCR-ABL mutation known as T315I has been recognized to cause resistance to all approved 1st and 2nd generation TKI.

More recently, a highly potent 3rd generation TKI called ponatinib has been developed and is the only approved TKI shown to be active against the T315I and all other resistance mutations. Initial studies combining ponatinib with chemotherapy have shown excellent response rates and promising survival in adult patients with newly diagnosed Ph+ ALL. However, in this group of patients ponatinib has not yet been directly compared with any of the other drugs, and there may be a moderately increased risk of vascular and cardiac adverse events, such as heart attacks, strokes or thrombosis.

Based on existing data, ponatinib shows great promise for treatment of Ph+ ALL, but its superiority over standard imatinib-based therapy in terms of long-term efficacy and safety need to be proven.

It is the main purpose of this trial to determine whether ponatinib is superior to imatinib when combined with the same chemotherapy that is considered a standard for elderly patients with Ph+ ALL. The study hypothesis is that a greater proportion of patients in the ponatinib arm will achieve a deep (molecular) response, and that survival without leukemia relapse will be superior. The side effects, safety and tolerability of the two treatment regimens will also be compared.

A second trial question will explore whether chemotherapy can be omitted from the treatment regimen by replacing it with an immunotherapy drug called blinatumomab. This is a type of antibody that activated the patient´s own immune cells (T-cells) and directs them to the leukaemia cells, which are then destroyed. This type of treatment has been very effective in patients with ALL that did not respond or returned after other types of therapy, and has been approved in the EU and USA as salvage therapy for ALL. By combining two very different types of targeted therapy, the TKI ponatinib and the antibody blinatumomab, we hope to deliver highly effective therapy for Ph+ ALL while eliminating the toxicity of chemotherapy.

To be able to compare these treatments, patients will be randomly assigned to the three treatment arms in a 1:1:1 ratio, i.e. the likelihood to be assigned to each of the treatment groups is the same. Overall duration of study treatment will be 2 years, followed by treatment with the TKI alone.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients > 55 years (biological age)
2. Philadelphia chromosome or BCR-ABL positive acute lymphoblastic leukaemia
3. Not previously treated except with corticosteroids, single dose vincristine or up to three doses of cyclophosphamide (maximum cumulative dose 1g/m2) or intrathecal therapy to control meningeal leukaemia
4. No uncontrolled CNS involvement
5. WHO performance status <2
6. Normal serum levels > LLN (lower limit of normal) of potassium and magnesium, or corrected to within normal limits with supplements, prior to the first dose of study medication
7. Signed written inform consent
8. Molecular evaluation for BCR-ABL1 performed
9. Willingness of sexually active male subjects whose sexual partners are women of childbearing potential (WOCBP), to use an effective form of contraception (pearl index < 1%) during the study and at least 6 months thereafter. Effective forms of contraception are complete sexual abstinence (refraining from heterosexual intercourse during the entire period of risk associated with the study treatments), combined oral contraceptive, hormone IUCD, vaginal hormone ring, transdermal contraceptive patch, contraceptive implant or depot contraceptive injection in combination with a second method of contraception like a condom or a cervical cap / diaphragm with spermicide or surgical sterilisation (vasectomy) in male patients.
10. Women of non-childbearing potential defined as sexually mature women who have undergone a hysterectomy or surgical sterilization or who have been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months).

Exclusion Criteria:

1. Patient previously treated with tyrosine kinase inhibitors
2. Known impaired cardiac function, including any of the following:

   * LVEF < 40%
   * Complete left bundle branch block
   * Right bundle branch block plus left anterior hemiblock, bifascicular block
   * History of or presence of clinically significant ventricular or atrial tachyarrhythmias
   * Clinically significant resting bradycardia (< 50 beats per minute)
   * Congenital long QT syndrome or QTcF >470 msec on screening ECG. If QTc > 470 msec and electrolytes are not within normal ranges before ponatinib dosing, electrolytes should be corrected and then the patient rescreened for QTcF criterion.
   * Myocardial infarction within 12 months prior to starting study treatment
   * Other clinical significant heart disease (e.g. unstable angina, congestive heart failure, uncontrolled hypertension)
3. Symptomatic peripheral vascular disease
4. Any history of ischemic stroke or transient ischemic attacks (TIAs)
5. Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention
6. History or presence of clinically relevant CNS pathology such as epilepsy, childhood or adult seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis (with exception of CNS leukemia that is well controlled with intrathecal therapy)
7. Active ALL in the CNS (confirmed by CSF analysis) or testes (by clinical assessment).
8. Autoimmune disease with potential CNS involvement
9. Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory) or active infection with Hepatitis B or C
10. Treatment with any other investigational agent or participating in another trial within 30 days prior to entering this study
11. Inadequate hepatic functions defined as ASAT or ALAT > 2,5 times the institutional upper limit of normal or > 5 times ULN if considered due to leukemia
12. Total bilirubin > 1.5-fold the institutional upper limit unless considered to be due to organ involvement by the leukemia or to M. Gilbert / M. Meulengracht
13. Concurrent severe diseases which exclude the administration of therapy
14. Chronic pancreatitis or acute pancreatitis as evidenced by clinical symptomatology and/or imaging within 6 months of study entry
15. Pregnant or lactating females
16. Patients unwilling or unable to comply with the protocol

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with a demonstrable molecular response | Within 5 months after start of study treatment
  Achievement of a molecular response in treatment arms 1 and 2 defined by a BCR-ABL1/ABL1 (B/A) transcript ratio of ≤10-4 by the time point scheduled for MRD analysis

IPD SHARING:
Plan to Share IPD: No
Access to data is subject to the standard operation procedures of the Sponsor, and requests for data will be reviewed accordingly. Data sharing is actively encouraged by accredited clinical trials units.